CLINICAL TRIAL: NCT07145931
Title: Tislelizumab Combined With Chemotherapy for Neoadjuvant Immunochemotherapy and Postoperative Adjuvant Therapy for Head and Neck Squamous Cell Carcinoma Invading the Skull Base: A Prospective, Single-arm, Phase II Clinical Study
Brief Title: Neoadjuvant Immunochemotherapy and Postoperative Adjuvant Immunotherapy for Head and Neck Squamous Cell Carcinoma Invading the Skull Base
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yujie Liang, MD, DDS, PhD, Associate Professor, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GHKQ-202503-L011
Record Dates: First submitted 2025-08-06; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer Squamous Cell Carcinoma; Skull Base--Cancer; Neoadjuvant Chemoimmunotherapy; Objective Response Rate
Keywords: Head and Neck Cancer Squamous Cell Carcinoma; Skull Base--Cancer; Neoadjuvant Chemoimmunotherapy; Objective response rate
MeSH Terms: interventions — Surgical Procedures, Operative; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): * Neoadjuvant therapy is administered every 3 weeks (Tislelizumab 200mg D1, Nab Paclitaxel 260mg/m² D1, Cisplatin 75mg/m² D1-3) for a total of 3 cycles.
  * Surgical treatment is performed within 3 weeks after completing neoadjuvant therapy.
  * Postoperative (chemo)radiotherapy is initiated 4-6 weeks after surgery.
  * Following (chemo)radiotherapy, adjuvant immunotherapy (Tislelizumab 200mg) is administered every 3 weeks for a total of 8 cycles.
  Interventions: Procedure: Neoadjuvant chemoimmunotherapy; Drug: Tislelizumab Nab paclitaxel

INTERVENTIONS:
Procedure: Neoadjuvant chemoimmunotherapy — * Neoadjuvant therapy is administered every 3 weeks (Tislelizumab 200mg D1, Nab Paclitaxel 260mg/m² D1, Cisplatin 75mg/m² D1-3) for a total of 3 cycles.
  * Surgical treatment is performed within 3 weeks after completing neoadjuvant therapy.
  * Postoperative (chemo)radiotherapy is initiated 4-6 weeks after surgery.
  * Following (chemo)radiotherapy, adjuvant immunotherapy (Tislelizumab 200mg) is administered every 3 weeks for a total of 8 cycles.
  Other Names: Surgery; Adjuvant immunotherapy
Drug: Tislelizumab Nab paclitaxel — Neoadjuvant therapy is administered every 3 weeks (Tislelizumab 200mg D1, Nab Paclitaxel 260mg/m² D1, Cisplatin 75mg/m² D1-3) for a total of 3 cycles.
  Other Names: Cisplatin

SUMMARY:
This prospective, single-arm, Phase II clinical trial aims to evaluate the efficacy and safety of tislelizumab combined with chemotherapy as neoadjuvant therapy and postoperative adjuvant immunotherapy in patients with skull base-invading head and neck squamous cell carcinoma. The primary objectives are to address the following questions:

* What are the objective response rate and pathological response of tislelizumab combined with chemotherapy as neoadjuvant therapy in patients with skull base-invading head and neck squamous cell carcinoma?
* Can neoadjuvant therapy convert unresectable skull base-invading head and neck squamous cell carcinoma into a resectable condition?
* Can adjuvant immunotherapy after neoadjuvant therapy prolong patients' recurrence-free survival and overall survival? The researchers will administer neoadjuvant therapy (tislelizumab combined with chemotherapy) and adjuvant immunotherapy to patients with skull base-invading head and neck squamous cell carcinoma and assess the treatment's efficacy and safety.

Participants will:

* Receive neoadjuvant therapy every 3 weeks (tislelizumab 200mg on Day 1, nab-paclitaxel 260mg/m² on Day 1, cisplatin 75mg/m² on Days 1-3) for 3 cycles.
* Undergo surgical treatment within 3 weeks after completing neoadjuvant therapy.
* Receive (chemo)radiotherapy 4-6 weeks after surgery.
* Receive adjuvant immunotherapy (tislelizumab 200mg) every 3 weeks after (chemo)radiotherapy for 8 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, regardless of gender;
* Histologically confirmed squamous cell carcinoma (including gingiva, buccal mucosa, palate, oropharynx, maxillary sinus, or maxilla/mandible) with radiological evidence of skull base invasion;
* Measurable tumor lesions (meeting RECIST v1.1 criteria);
* Treatment-naïve primary T4b-stage patients (N any, per AJCC 8th Edition, 2017);
* ECOG PS score: 0-1;
* Medically fit for surgery and chemotherapy, with no surgical contraindications;
* Women of childbearing potential (18-49 years) must have a negative pregnancy test within 7 days before treatment. Sexually active men and women must agree to use effective contraception during the trial and for 3 months after treatment cessation;
* Willing to provide written informed consent and comply with scheduled follow-ups, treatments, lab tests, and other study requirements.

Exclusion Criteria:

* Previous anti-tumor treatments including chemotherapy, radiotherapy, or immunotherapy; Refusal to sign informed consent;
* Patients who refuse the study treatment protocol; patients unable to complete treatment as planned; or patients unable to comply with regular follow-up due to psychological, social, familial or geographical reasons;
* Patients with known allergies to any study medications;
* Patients with poor systemic conditions unfit for treatment: as determined by routine tests (complete blood count, blood biochemistry, ECG, chest X-ray, etc.). Poor systemic conditions include: hemoglobin <60g/L, WBC <3.0×10⁹/L, platelets <80×10⁹/L, or serum creatinine >133μmol/L - such patients may be recommended for conservative treatment;
* Patients with autoimmune diseases requiring long-term immunosuppressive or corticosteroid therapy;
* Pregnant or lactating women (pregnancy testing should be considered for sexually active women of childbearing potential);
* Patients with current or previous malignancies (except adequately treated non-melanoma skin cancer, cervical carcinoma in situ, or papillary thyroid carcinoma);
* Participation in other clinical trials within 30 days prior to enrollment;
* Other conditions that may compromise patient safety or compliance as assessed by investigators, including: severe comorbidities (including psychiatric disorders), significantly abnormal laboratory results, or other high-risk familial/social factors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2027-09-20 (Estimated); Study Completion 2029-09-20 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Within 3 weeks after completion of neoadjuvant therapy
  Objective Response Rate (ORR) is a pivotal efficacy endpoint in oncology therapeutic evaluation, defined as the proportion of patients whose tumor burden shrinks to a prespecified threshold (achieving either complete or partial response). This metric is measured using internationally standardized criteria (RECIST 1.1), with radiographic imaging to monitor changes in the sum of target lesion diameters. Based on Standardized Criteria (e.g., RECIST 1.1). Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): ≥30% decrease in tumor size (sum of target lesions). ORR = CR + PR (expressed as a percentage).

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Until 21 days after the end of the study
  To evaluate the adverse events during the study period according to the NCI-CTCAE, version 5.0, including vital signs, physical examination, laboratory tests, changes in ECOG score, etc., as well as adverse events and serious adverse events, are calculated to the incidence of adverse events and serious adverse events.
Pathologic Efficacy | Perioperative
  The percentage of residual tumor cells in tumor bed of pathological specimens after surgery. Pathological complete response (pCR) refers to tumors the absence of any viable tumor cells within the tumor bed. Major pathological response (MPR) is defined as 10% or fewer residual viable tumor cells within the tumor bed.
Clinical Downstaging Rate | Within 3 weeks after completion of neoadjuvant therapy.
  The proportion of patients with reduction in clinical TNM stage.
Surgical Conversion Rate | Within 3 weeks after completion of neoadjuvant therapy.
  The proportion of patients with initially unresectable tumors that become resectable after treatment.
R0 Resection Rate | Perioperative
  The proportion of patients achieving complete tumor removal with microscopically negative margins (no residual tumor cells).
Organ Preservation Rate | Perioperative
  The proportion of patients who, despite pretreatment tumor invasion into critical organs (e.g., eyeball, internal carotid artery, dura mater), successfully retain the involved organ while still achieving R0 resection.
Recurrence-Free Survival | Until cancer recurrence or death or the last follow-up, whichever came first, assessed up to 24 months
  The time from enrollment until cancer recurrence or death from any cause.
Overall Survival | Until death from any cause or the last follow-up, whichever came first, assessed up to 24 months
  The time from enrollment until death from any cause or the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Liang, Principal Investigator — Hospital of Stomatology, Sun Yat-Sen University
Locations (1):
- Hospital of Stomatology, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 6 months after publication
Access Criteria: The researchers obtained study protocol, statistical analysis plan, informed consent form, clinical study report, analytic code via email communication.

REFERENCES:
- [Background] Zhang Z, Wu B, Peng G, Xiao G, Huang J, Ding Q, Yang C, Xiong X, Ma H, Shi L, Yang J, Hong X, Wei J, Qin Y, Wan C, Zhong Y, Zhou Y, Zhao X, Leng Y, Zhang T, Wu G, Yao M, Zhang X, Yang K. Neoadjuvant Chemoimmunotherapy for the Treatment of Locally Advanced Head and Neck Squamous Cell Carcinoma: A Single-Arm Phase 2 Clinical Trial. Clin Cancer Res. 2022 Aug 2;28(15):3268-3276. doi: 10.1158/1078-0432.CCR-22-0666. PMID 35766967
- [Background] Patel SA, Gibson MK, Deal A, Sheth S, Heiling H, Johnson SM, Douglas K, Flores M, Blumberg J, Lumley C, Yarbrough WG, Shen C, Chera BS, Bauman JR, Hackman T, Weiss J. A phase 2 study of neoadjuvant chemotherapy plus durvalumab in resectable locally advanced head and neck squamous cell carcinoma. Cancer. 2023 Nov 1;129(21):3381-3389. doi: 10.1002/cncr.34930. Epub 2023 Jul 3. PMID 37395170
- [Background] Wu D, Li Y, Xu P, Fang Q, Cao F, Lin H, Li Y, Su Y, Lu L, Chen L, Li Y, Zhao Z, Hong X, Li G, Tian Y, Sun J, Yan H, Fan Y, Zhang X, Li Z, Liu X. Neoadjuvant chemo-immunotherapy with camrelizumab plus nab-paclitaxel and cisplatin in resectable locally advanced squamous cell carcinoma of the head and neck: a pilot phase II trial. Nat Commun. 2024 Mar 11;15(1):2177. doi: 10.1038/s41467-024-46444-z. PMID 38467604
- [Background] Zhong LP, Zhang CP, Ren GX, Guo W, William WN Jr, Sun J, Zhu HG, Tu WY, Li J, Cai YL, Wang LZ, Fan XD, Wang ZH, Hu YJ, Ji T, Yang WJ, Ye WM, Li J, He Y, Wang YA, Xu LQ, Wang BS, Kies MS, Lee JJ, Myers JN, Zhang ZY. Randomized phase III trial of induction chemotherapy with docetaxel, cisplatin, and fluorouracil followed by surgery versus up-front surgery in locally advanced resectable oral squamous cell carcinoma. J Clin Oncol. 2013 Feb 20;31(6):744-51. doi: 10.1200/JCO.2012.43.8820. Epub 2012 Nov 5. PMID 23129742
- [Background] Sharma P, Stecklein SR, Yoder R, Staley JM, Schwensen K, O'Dea A, Nye L, Satelli D, Crane G, Madan R, O'Neil MF, Wagner J, Larson KE, Balanoff C, Kilgore L, Phadnis MA, Godwin AK, Salgado R, Khan QJ, O'Shaughnessy J. Clinical and Biomarker Findings of Neoadjuvant Pembrolizumab and Carboplatin Plus Docetaxel in Triple-Negative Breast Cancer: NeoPACT Phase 2 Clinical Trial. JAMA Oncol. 2024 Feb 1;10(2):227-235. doi: 10.1001/jamaoncol.2023.5033. PMID 37991778
- [Background] Romero D. Neoadjuvant chemoimmunotherapy is effective in locally advanced cervical cancer. Nat Rev Clin Oncol. 2024 Feb;21(2):84. doi: 10.1038/s41571-023-00855-x. No abstract available. PMID 38110599
- [Background] Sepesi B, Swisher SG. Role of neoadjuvant chemoimmunotherapy for resectable NSCLC. Nat Rev Clin Oncol. 2022 Aug;19(8):497-498. doi: 10.1038/s41571-022-00647-9. No abstract available. PMID 35585121
- [Background] Masarwy R, Kampel L, Horowitz G, Gutfeld O, Muhanna N. Neoadjuvant PD-1/PD-L1 Inhibitors for Resectable Head and Neck Cancer: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2021 Oct 1;147(10):871-878. doi: 10.1001/jamaoto.2021.2191. PMID 34473219
- [Background] Burtness B, Harrington KJ, Greil R, Soulieres D, Tahara M, de Castro G Jr, Psyrri A, Baste N, Neupane P, Bratland A, Fuereder T, Hughes BGM, Mesia R, Ngamphaiboon N, Rordorf T, Wan Ishak WZ, Hong RL, Gonzalez Mendoza R, Roy A, Zhang Y, Gumuscu B, Cheng JD, Jin F, Rischin D; KEYNOTE-048 Investigators. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019 Nov 23;394(10212):1915-1928. doi: 10.1016/S0140-6736(19)32591-7. Epub 2019 Nov 1. PMID 31679945
- [Background] Cohen EEW, Soulieres D, Le Tourneau C, Dinis J, Licitra L, Ahn MJ, Soria A, Machiels JP, Mach N, Mehra R, Burtness B, Zhang P, Cheng J, Swaby RF, Harrington KJ; KEYNOTE-040 investigators. Pembrolizumab versus methotrexate, docetaxel, or cetuximab for recurrent or metastatic head-and-neck squamous cell carcinoma (KEYNOTE-040): a randomised, open-label, phase 3 study. Lancet. 2019 Jan 12;393(10167):156-167. doi: 10.1016/S0140-6736(18)31999-8. Epub 2018 Nov 30. PMID 30509740
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Argiris A, Karamouzis MV, Raben D, Ferris RL. Head and neck cancer. Lancet. 2008 May 17;371(9625):1695-709. doi: 10.1016/S0140-6736(08)60728-X. PMID 18486742
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Ganly I, Patel SG, Singh B, Kraus DH, Bridger PG, Cantu G, Cheesman A, De Sa G, Donald P, Fliss DM, Gullane P, Janecka I, Kamata SE, Kowalski LP, Levine PA, Medina Dos Santos LR, Pradhan S, Schramm V, Snyderman C, Wei WI, Shah JP. Craniofacial resection for malignant paranasal sinus tumors: Report of an International Collaborative Study. Head Neck. 2005 Jul;27(7):575-84. doi: 10.1002/hed.20165. PMID 15825201
- [Background] Head and neck squamous cell carcinoma. Nat Rev Dis Primers. 2020 Nov 26;6(1):93. doi: 10.1038/s41572-020-00233-2. No abstract available. PMID 33243985